CLINICAL TRIAL: NCT01193621
Title: Early Clinical Evaluation of the Pharmacokinetics and Mechanism Based Pharmacodynamics of Haloperidol Using Positron Emission Tomography in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Kyun-Seop Bae, Associate Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 2009-0692
Record Dates: First submitted 2010-09-01; First posted 2010-09-02 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-07

CONDITIONS: Healthy
Keywords: early evaluation; pharmacokinetics; pharmacodynamics; Biodistribution; D2-receptor occupancy
MeSH Terms: interventions — Haloperidol; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- haloperidol (Active Comparator): 0.5, 1, 3 mg of haloperidol will be administered orally every 24 hours for 7 days to 4 healthy subjects in each dose level (a total of 12 subjects).
  Dose groups are as follows; D2-receptor occupancy study Group Single Oral Dose No. of subjects
  1. 0.5 mg 4
  2. 1 mg 4
  3. 5 mg 4
  Interventions: Drug: haloperidol, PET

INTERVENTIONS:
Drug: haloperidol, PET — 1. Biodistribution study Intravenous 18F haloperidol(10 mCi) Dose injection two times before whole body PET scan
  2. D2-receptor occupancy study Group Doses No. of subjects 1 0.5 mg 4 2 1 mg 4 3 3 mg 4
  above doses will be administrated orally every 24 hours for 7 days.

SUMMARY:
In the present study, the investigators will establish the clinical trial technology for early evaluation of drug characteristics in terms of pharmacokinetics and pharmacodynamics for haloperidol as a model drug, using positron emission tomography.

DETAILED DESCRIPTION:
1. Study Design

   This study will consist of two parts. One is "biodistribution study of haloperidol" in 12 subjects, and the other is "receptor occupancy study of haloperidol" in 12 subjects. In the biodistribution study, 18F-haloperidol (10 mCi) will be injected intravenously two times into each of the 12 subjects (cross-over design). Whole body PET will be conducted after the first haloperidol injection and local brain PET after the 2nd haloperidol injection after the 7 day washout period.

   1.1 D2-receptor occupancy study Group Doses No. of subjects 1 0.5 mg 4 2 1 mg 4 3 3 mg 4
2. Measurement 2.1 The D2 receptor Occupancy of haloperidol.
3. Test schedule 3.1 Biodistribution study

   * Whole body PET (day 1)
   * Brain local PET (day 8) 3.2 Receptor occupancy study
   * Baseline PET before drug administration (day 1 0h), 6h (day 1 6h), 24h (day 2 0h), after the first haloperidol administration (day 1 0h), and 24 h (day 8), 72 h (day 10), and 168 h (day 14) after the last dosing of haloperidol (day 7 0h).
   * Drug administration from day 1 through day 7 every 24 hours PK blood sampling (6 ml, each) prior to the first haloperidol administration (day 1 0h) and 6h (1 day 6h), 24h (2 day 0h), 48 h (3 day 0h), 96 h (5 day 0h), 144 h (7 day 0h) and, 0.5, 1, 2, 4, 6, 8, 12, 24 h (8day 0h), 48h (9day 0h), 72h (10 day 0h) after taking the last oral dose of haloperidol
4. Analytic Methods 4.1 Pharmacokinetics: Noncompartmental Analysis Using Winnonlin Compartment model using NONMEM VII 4.2 Pharmacodynamics in the brain: Emax or linear model using NONMEM VII

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy males as determined by medical history and physical examination
* Age from 19 to 45 years
* Weight ≥ 45 kg and within ± 20% of IBW
* Clinical laboratory test results within normal reference range for the National Cancer Center, Hospital or results with minor deviations which are judged to be not clinically significant by the investigator
* Normal blood pressure and heart rate (supine and standing) as determined by the investigator
* Are reliable and willing to make themselves available for the duration of the study, and who will abide by the study restrictions
* Have given written informed consent

Exclusion Criteria:

* History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, neurological disorders capable of altering the absorption, metabolism or elimination of drugs, or of constituting a risk factor when taking the study medication
* An episode of febrile disease or infectious disease within the past 2 weeks
* Evidence of significant active hematologic disease and/or blood donation in the last 2 months
* Evidence of significant active neuropsychiatric disease
* Regular use of drugs or abuse
* History of drug hypersensitivity or clinically significant allergic reactions of any origin
* Participation in a study involving administration of an investigational compound within the past 30 days
* Have a regular alcohol intake greater than 21 units/week or subjects unwilling to stop alcohol for the duration of the study periods
* Intend to use concomitant drug therapy, including non prescription medication on a regular basis apart from vitamin/mineral supplements
* Smoking history for recent 3 months
* Use of medication within 7 days prior to the study. If this situation arises inclusion of an otherwise suitable volunteer may be at the discretion of the investigator

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2008-01; Primary Completion 2010-07 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
plasma haloperidol concentration | day 1 0h (predose), day 1 6h, day 2 0h, day 3 0h (predose), day 5 0h (predose), and day 7 0h (predose), 0.5, 1, 2, 4, 6, 8, 12, 24(day 8 0h), 48(day 9 0h), 72h (day 10h)

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, Seoul, South Korea